CLINICAL TRIAL: NCT06458998
Title: Getting To Implementation: Comparing the Effectiveness of Implementation Strategies to Improve Cancer Screening for Veterans
Brief Title: Getting To Implementation: Improving Cancer Screening for Veterans
Acronym: GTI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Shari Rogal, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24010054; 1792560 (Other: VA Pittsburgh Healthcare System); BPS-2023C1-31034 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cancer of Liver; Cancer of Colon; Cirrhosis
Keywords: implementation strategies; patient navigation; implementation facilitation; Consolidated Framework for Implementation Research; Early detection of cancer
MeSH Terms: conditions — Liver Neoplasms; Colonic Neoplasms; Fibrosis | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Navigation (PN) (Active Comparator): Half of the HCC sites and half of the CRC sites will be randomized to PN delivered by Clinical Resource Hub navigators.
  Interventions: Behavioral: Patient Navigation
- Implementation Facilitation (IF) (Active Comparator): Half of the HCC sites and half of the CRC sites will be randomized to IF delivered by 2 facilitators (one clinical and one evaluation expert) per site.
  Interventions: Behavioral: Implementation Facilitation

INTERVENTIONS:
Behavioral: Patient Navigation — Clinical Resource Hub (CRH) providers include a small group of nurses, advance practice providers, and physicians who work to improve care across a range of measures using virtual PN. CRH providers will 1) use existing dashboards to identify at-risk Veterans, 2) conduct Veteran outreach (two calls, one letter) to provide education, problem solve, and offer screening, 3) order and schedule HCC or CRC screening tests, and 4) provide reminders and follow up on results.
  Arms: Patient Navigation (PN)
Behavioral: Implementation Facilitation — Facilitators will provide 20 hours of virtual facilitation to site teams, through 1-hour meetings every other week and ad hoc meetings, over 12 months. They will guide site teams through a seven-step playbook called Getting To Implementation (GTI), which uses a series of tools to select context-specific strategies.
  Arms: Implementation Facilitation (IF)

SUMMARY:
Gastrointestinal cancers such as colon cancer and liver cancer cause many deaths in the US. Testing could catch these cancers early, helping people live longer. The goal of this study is to compare two different ways of getting more people tested for these cancers: 1) by directly reaching out to the people who need testing or 2) by helping providers fix issues that hold up testing.

The main question it aims to answer is: how should healthcare systems go about choosing one or the other?

Researchers will look at cancer testing rates over time at sites that are trying these different approaches. They will also survey and interview participants from these sites.

DETAILED DESCRIPTION:
Researchers will conduct two hybrid type 3, cluster-randomized trials to compare the effectiveness of Patient Navigation (PN) and Implementation Facilitation (IF) on hepatocellular cancer (HCC) and colorectal cancer (CRC) screening completion. Trials will enroll 24 sites for the HCC arm and 32 sites for the CRC arm, passively enrolling and cluster-randomizing Veterans by their site of primary care. Multi-level implementation determinants (i.e., barriers and facilitators), preconditions, and moderators will also be evaluated pre- and post-intervention, using Consolidated Framework for Implementation Research (CFIR)-mapped surveys and interviews of Veteran participants and provider participants. Comparing findings in the two trials will allow researchers to understand how the barriers and strategies operate differently for a one-time screening in a relatively healthy population (CRC) vs. repeated screening in a more medically complex population (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Veterans:

   * ≥18 years of age
   * Enrolled in Veterans Health Administration (VA)
   * Have ≥1 VA encounter in the prior 18 months
   * Hepatocellular cancer (HCC) screening subgroup: Diagnosis of cirrhosis in electronic medical record
   * Colorectal cancer (CRC) screening subgroup: ≥45 years of age, positive fecal immunochemical test (FIT) (or other screening stool test) in the last 18 months
2. Providers:

   * Healthcare provider or related staff at participating VA site or engaged in CRC or HCC screening pathways in an included VA site (e.g., scheduling)
   * ≥18 years of age

Exclusion Criteria:

1. Veterans:

   * <18 years of age
   * Not enrolled in VA
   * No VA encounters in the prior 18 months
   * Limited life expectancy (< 6 months), defined as having a code for hospice
2. Providers:

   * Members of the study team will not participate, even if their sites are recruited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30300 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Reach of HCC screening from Baseline to 12 months | Baseline, 12 months from Baseline
  Reach of an intervention refers to the absolute number, proportion, and representativeness of individuals who are willing to participate in a given intervention. The reach outcome will be the percentage of eligible Veterans in the HCC screening subgroup receiving guideline-concordant abdominal imaging within the prior 6 months.
Change in Reach of CRC screening from Baseline to 12 months | Baseline, 12 months from Baseline
  Reach of an intervention refers to the absolute number, proportion, and representativeness of individuals who are willing to participate in a given intervention. The reach outcome will be the percentage of eligible Veterans in the CRC screening subgroup receiving a colonoscopy.

SECONDARY OUTCOMES:
Effectiveness of screening - Change in the number of tumor/polyp/lesions detected from Baseline to 12 months | Baseline, 12 months from Baseline
  Effectiveness is the impact of an intervention on important individual outcomes, defined as detection of cancer.
Effectiveness of screening - Change in time to treatment from Baseline to 12 months | Baseline, 12 months from Baseline
  Effectiveness is the impact of an intervention on important individual outcomes, defined as time to treatment, which will be measured from the date of cancer diagnosis to the date of referral.
Change in Adoption of screening from Baseline to 12 months | Baseline, 12 months from Baseline
  Adoption is the absolute number, proportion, and representativeness of settings/people who are willing to initiate a program. Site-level adoption will be defined as meeting the national goal of 65% HCC screening and 80% linkage to colonoscopy within 6-months of positive stool-based screening.
Feasibility of intervention assessed by the Feasibility of Intervention measure (FIM) | 12 months from Baseline
  Feasibility refers to the extent to which an intervention can be successfully used within a given setting, as measured by the Feasibility of Intervention Measure (FIM) assessment. The FIM is a 4-item measure, with each item scored using a 5-point Likert scale. Scores range from a minimum of 4 points to a maximum of 20. Higher scores indicate greater feasibility.
Acceptability assessed by the Acceptability of Intervention Measure (AIM) | 12 months from Baseline
  Acceptability refers to a given intervention being perceived as agreeable, palatable, or satisfactory by implementation stakeholders, as measured by the Acceptability of Intervention Measure (AIM). The AIM is a 4-item measure, with each item scored using a 5-point Likert scale. Scores range from a minimum of 4 points to a maximum of 20. Higher scores indicate greater acceptability.
Appropriateness assessed by the Intervention Appropriateness Measure (IAM) | 12 months from Baseline
  Appropriateness is the perceived fit of an intervention to address a particular issue or problem, as measured by the Intervention Appropriateness Measure (IAM). The IAM is a 4-item measure, with each item scored using a 5-point Likert scale. Scores range from a minimum of 4 points to a maximum of 20. Higher scores indicate greater appropriateness.
Fidelity - Proportion of Veterans receiving recommended screening | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Fidelity is the degree to which an intervention/innovation is delivered as intended. Fidelity of cancer screenings will be assessed by the proportion of Veterans at a given site receiving HCC or CRC screening as recommended (correct timing and modality). Fidelity to core strategy elements will be evaluated using checklists.
Maintenance of HCC Screening at 18 and 24 months from Baseline | 6 months post-intervention (18 months from Baseline), 12 months post-intervention (24 months from Baseline)
  Maintenance is the extent to which a program becomes part of routine organizational practices. Sustainment of HCC Screening will be measured by the percentage of eligible Veterans in the HCC screening subgroup receiving guideline-concordant abdominal imaging within the prior 6 months.
Maintenance of CRC Screening at 18 and 24 months from Baseline | 6 months post-intervention (18 months from Baseline), 12 months post-intervention (24 months from Baseline)
  Maintenance is the extent to which a program becomes part of routine organizational practices. Sustainment of CRC Screening will be measured by the percentage of eligible Veterans in the CRC screening subgroup receiving a colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Shari S Rogal, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogal SS, Yakovchenko V, Morgan TR, Dominitz JA, McCurdy H, Nobbe A, Ekanem NR, Kang C, Gonzalez RI, Park A, Anwar J, Neely B, Gibson S, Lamorte C, Bajaj JS, Patton HM, Yao Y, Gawron AJ. Comparing the effectiveness of implementation strategies to improve liver and colon cancer screening for Veterans: protocol for a large cluster-randomized implementation study. Implement Sci. 2025 Aug 9;20(1):38. doi: 10.1186/s13012-025-01448-1. PMID 40783525